CLINICAL TRIAL: NCT01506011
Title: An Open-label Randomized, Single Dose, Two Way Crossover Oral Bioequivalence Study of Amlodipine Besylate/Benazepril HCl Capsules of Dr. Reddy's With Lotrel® Capsules of Novartis in Human Subjects Under Fasting Conditions.
Brief Title: Bioequivalence Study of Amlodipine Besylate/Benazepril HCl 10 mg/40 mg Capsules of Dr. Reddy's Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 5530/06-07
Record Dates: First submitted 2012-01-05; First posted 2012-01-09 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting | interventions — benazepril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amlodipine Besylate/Benazepril HCl (Experimental): Amlodipine Besylate/Benazepril HCl 10 mg/40 mg capsules of Dr. Reddy's Laboratories Ltd.
  Interventions: Drug: Amlodipine Besylate/Benazepril HCl
- Lotrel (Active Comparator): Lotrel® Amlodipine Besylate/Benazepril HCl 10 mg/40 mg capsules of Novartis Pharmaceuticals
  Interventions: Drug: Amlodipine Besylate/Benazepril HCl

INTERVENTIONS:
Drug: Amlodipine Besylate/Benazepril HCl — Amlodipine Besylate/Benazepril HCl 10 mg/40 mg capsules
  Other Names: Lotrel

SUMMARY:
The purpose of this study single dose bioequivalence of Amlodipine Besylate/Benazepril HCl 10 mg/40 mg capsules with Lotrel® capsules in healthy human subjects and monitor clinical status, adverse events and laboratory investigations and assess relative safety and tolerance under fasting conditions

DETAILED DESCRIPTION:
An open-label randomized, single dose, two way crossover oral bioequivalence study to compare Amlodipine Besylate/Benazepril Hydrochloride 10 mg/40 mg capsules (Dr. Reddy's Laboratories Ltd.,) with Lotrel® capsules Novartis Pharmaceuticals Corporation in healthy human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will provide written informed consent.
* Subjects must be healthy adults within 18-45 years of age (inclusive).
* Body mass index of ≥18 kg/m2 and ≤25 kg/m2, with body weight not less than 50 kg.
* Subjects must be of normal health as determined by medical history and physical examination performed within 15 days prior to the dosing of period I.
* Have normal ECG, Chest X-ray and vital signs.
* Availability of subject for the entire study period and willingness to adhere to protocol requirements as evidenced by written informed consent.
* If subject is a female volunteer and is of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device(IUD), or abstinence.

or is postmenopausal for at least 1 year. or is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject)

•Each female subject will be given a urine pregnancy test at check-in for period-I, period-II and post study.

Exclusion Criteria:

* Subjects incapable of understanding the informed consent.
* Subjects with BP ≤90/60 mm/Hg or BP ≥140/90 mm/Hg
* History of hypersensitivity or idiosyncratic reaction to Amlodipine Besylate/Benazepril Hydrochloride or any other related drug.
* Any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal function. Subjects with a history of tuberculosis, epilepsy, asthma(during past 5 years),diabetes, psychosis or glaucoma will not be eligible for the study
* Regular smoker who smokes more than ten cigarettes daily and has difficulty in abstaining from smoking for the duration of each study period.
* Subjects who has taken over the counter or prescribed medications, including any enzyme modifying drugs or any systemic medication within the past 30 days prior to dosing in Period-I.
* History of any psychiatric illness, which may impair the ability to provide written, informed consent.
* Subjects who have a history of alcohol or substance abuse within the last 5 years
* Subjects with clinically significant abnormal values of laboratory parameters.
* Subjects who have participated in any other clinical investigation using experimental drug or had bled more than 350 mL in the past 3 months.
* Subjects who are unable to or likely to be non-compliant with protocol requirements or restrictions.
* Any subject in whom Amlodipine Besylate /Benazepril Hydrochloride is contraindicated for medical reasons
* Subjects who are intolerant to venipuncture
* Subjects with positive urine screen for drugs of abuse. All subjects will have urine samples assayed for the presence of drugs of abuse as part of the clinical laboratory screening procedures and at each study period check-in. Subjects found to have urine concentrations of any of the tested drugs will not be allowed to participate
* Female volunteers who has used implanted or injected hormonal contraceptives anytime during the 6 months prior to study or used hormonal contraceptives within 14 days before dosing
* Female volunteers demonstrating a positive pregnancy screen.
* All female subjects will be screened for pregnancy at check-in each study period. Subjects with positive or inconclusive results will be withdrawn from the study
* Female volunteers who are currently breast feeding.
* Female subjects who are pregnant, breast-feeding, or who are likely to become pregnant during the study will not be allowed to participate. Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable barrier method (e.g. condom, IUD) of contraception during the course of the study (first dosing until last blood collection) or they will not be allowed to participate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2007-03; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence is based on Cmax and AUC parameters | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: I. S. Gandhi., MD, Principal Investigator — Vimta Labs Ltd.
Locations (1):
- Vimta Labs Ltd., Hyderabad, A.P, India